CLINICAL TRIAL: NCT06990776
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQA3605 Tablets in Treatment-naive HBeAg-positive Subjects With Chronic HBV Infection
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of TQA3605 Tablets in Treatment-naive Chronic HBV-infected Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Per sponsor request. Premature closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQA3605-II-02
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 100mg TQA3605 tablets + entecavir (ETV) (PART A) (Experimental): Patients aged 30-65 years old group：TQA3605 tablets, 100mg once a day, orally for 48 weeks in combination with entecavir, followed by treatment with entecavir for 24 weeks
  Interventions: Drug: TQA3605 Tablets; Drug: Entecavir dispersible tablets
- 200mg TQA3605 tablets +ETV (PART A) (Experimental): Patients aged 30-65 years old group：TQA3605 tablets, 200mg once a day, orally for 48 weeks in combination with entecavir, followed by treatment with entecavir for 24 weeks
  Interventions: Drug: TQA3605 Tablets; Drug: Entecavir dispersible tablets
- TQA3605 tablets Placebo +ETV (PART A) (Placebo Comparator): Patients aged 30-65 years old group： TQA3605 tablets placebo, once a day, orally for 48 weeks in combination with entecavir, followed by treatment with entecavir for 24 weeks.
  Interventions: Drug: TQA3605 tablets Placebo
- 200mg TQA3605 tablets +ETV (PART B) (Experimental): Patients aged 18-30 years old group：TQA3605 tablets, 200mg once a day, orally for 48 weeks in combination with entecavir, followed by treatment with entecavir for 24 weeks.
  Interventions: Drug: TQA3605 Tablets; Drug: Entecavir dispersible tablets
- TQA3605 tablets Placebo +ETV (PART B) (Placebo Comparator): Patients aged 18-30 years old group：TQA3605 tablets Placebo taken once a day, orally for 48 weeks in combination with entecavir, followed by treatment with entecavir for 24 weeks.
  Interventions: Drug: TQA3605 tablets Placebo

INTERVENTIONS:
Drug: TQA3605 tablets Placebo — Placebo contains no active substance.
  Arms: TQA3605 tablets Placebo +ETV (PART A); TQA3605 tablets Placebo +ETV (PART B)
Drug: TQA3605 Tablets — TQA3605 tablets is core protein allosteric modulators
  Arms: 100mg TQA3605 tablets + entecavir (ETV) (PART A); 200mg TQA3605 tablets +ETV (PART A); 200mg TQA3605 tablets +ETV (PART B)
Drug: Entecavir dispersible tablets — Entecavir dispersible tablets is an inhibitor of hepatitis B virus replication.
  Arms: 100mg TQA3605 tablets + entecavir (ETV) (PART A); 200mg TQA3605 tablets +ETV (PART A); 200mg TQA3605 tablets +ETV (PART B)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase II study, in which all participants are required to use TQA3605 tablets/placebo in combination with entecavir. The purpose is to evaluate the efficacy and safety of TQA3605 tablets combined with entecavir in treatment-naive chronic HBV-infected subjects. A total of 215 subjects are required.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old (including boundary values), regardless of gender;
* Screening requires virological , clinical or pathological evidence of hepatitis B virus infection for more than 6 months; HBsAg positive, HBeAg positive, ALT≤5×ULN at screening;
* Never received nucleoside (acid) analog or interferon treatment, or previously received no more than 12 weeks of treatment but had discontinued therapy at least 6 months prior to the screening visit;
* Ability to communicate effectively with researchers and understand and comply with the requirements of this study, understand and sign the informed consent form;
* Male subjects with female partners who have fertility or female subjects of childbearing age are willing to voluntarily adopt effective contraceptive measures screening to within 3 months after leaving the group.

Exclusion Criteria:

* Pregnant (positive pregnancy test) or lactating women.
* Co-infection with other viruses such as Hepatitis A Virus (HAV), Hepatitis C Virus (HCV), Hepatitis D Virus (HDV), Hepatitis E Virus (HEV), Human Immunodeficiency Virus (HIV), Syphilis, etc.;
* History of cirrhosis or evidence of significant fibrosis or cirrhosis before or during screening;
* History of hepatocellular carcinoma (HCC) or suspected HCC before or during screening.;
* History of malignant tumors within the past 5 years prior to screening, except for certain cancers that can be completely cured by surgical resection;
* Subjects with other chronic liver diseases, including but not limited to autoimmune liver disease, alcoholic liver disease, Wilson's disease, Gilbert syndrome, etc;
* Previous organ or bone marrow transplantation;
* Clinically significant abnormal laboratory test results at screening.
* Poorly controlled thyroid diseases or clinically significant thyroid dysfunction;
* Autoimmune diseases;
* Significant systemic or major illnesses other than liver disease.
* Any systemic anti-tumor or immunosuppressive therapy, or immunomodulatory therapy within 6 months prior to screening.
* High-dose systemic corticosteroids use within 3 months prior to screening;
* History of alcohol or drug abuse within the past year or excessive alcohol consumption.
* History of blood transfusion within 2 months prior to screening;
* History of allergy to investigational drug or its excipients.
* Previously participated in the clinical trial of hepatitis B core protein allosteric modulators;
* Participation in another clinical trial and receipt of an investigational drug within the following timeframes before the first dose in this study: 5 half-lives (if known) or twice the duration of the biological effect of the study treatment (if known), whichever is longer, or 90 days (if the half-life or duration is unknown);
* History or condition of cardiovascular disease;
* Any other condition deemed inappropriate for inclusion by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
hepatitis B virus (HBV) DNA <10 IU/mL | 48 weeks
  Percentage of subjects with HBV DNA below the lower limit of quantification (<10 IU/mL) after 48 weeks of treatment.

SECONDARY OUTCOMES:
Percentage of subjects with HBV DNA<10 IU/mL | 12 weeks, 24 weeks, 36 weeks, 60 weeks, 72 weeks
  Percentage of subjects with HBV DNA<10 IU/mL at week 12, 24, 36, 60, and 72
Percentage of HBV DNA<20 IU/mL | 12 weeks, 24 weeks, 36 weeks, 48weeks, 60 weeks, 72 weeks
  Percentage of subjects with HBV DNA<20 IU/mL at weeks 12, 24, 36, 48, 60, and 72 of treatment.
Percentage of subjects with HBeAg serologic clearance and/or serologic conversion | 24weeks, 48 weeks, 72 weeks
  Percentage of subjects with HBeAg serologic clearance and/or serologic conversion
Alanine aminotransferase(ALT)≤The upper limit of the normal reference value (ULN) | 24weeks, 48 weeks, 72 weeks
  The rate of ALT normalization at weeks 24, 48, and 72 of treatment
Virology breakthrough percentage | 24weeks, 48 weeks, 72 weeks
  Percentage of subjects who experienced virological breakthroughs at weeks 24, 48, and 72 of treatment
Actual values of HBV markers and changes over time relative to baseline | 12 weeks, 24 weeks, 36 weeks, 48 weeks, 72 weeks
  Actual values of HBsAg, HBeAg, HBV DNA, HBV RNA, and Hepatitis B core-related antigen (HBcrAg) at each visit time point and their changes over time relative to baseline.
Adverse events (AE) | 72 weeks
  The incidence and severity of adverse events.
Steady state minimum concentration (Cmin,ss) | 48 weeks
  Cmin,ss of TQA3605 and its metabolite

CONTACTS AND LOCATIONS:
Locations (29):
- China (29):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Southwest Hospital of AMU, Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - NanFang Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of GUANGXI Medical University, Nanning, Guangxi
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Zhengzhou No.6 peoples Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Hospital of Changsha, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Naniing Drum Tower Hospital, Nanjing, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - The Fifth People's Hospital of Wuxi, Wuxi, Jiangsu
  - Zhenjiang Third People's Hospital, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Xi'an Jiaotong University Second Affiliated Hospital, Xi'an, Shaanxi
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Clinical Center for Public Health, Jinan, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yiwu Central Hospital, Yiwu, Zhejiang